CLINICAL TRIAL: NCT00050063
Title: A Rollover Study of A5058s: A Phase II Trial to Evaluate the Ability of Vaccine-Induced Helper and CTL Responses to Control Viremia in the Absence of Antiretroviral Therapy
Brief Title: Effects of Therapeutic HIV Vaccination on Control of HIV After Discontinuation of Anti-HIV Drugs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: A5172; 10184 (Registry Identifier: DAIDS ES Registry Number); ACTG A5172
Record Dates: First submitted 2002-11-20; First posted 2002-11-21 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Therapeutic Vaccine; Treatment Experienced; AIDS Vaccines; Treatment Interruption; Viral Load; T-Lymphocytes, Cytotoxic; T-Lymphocytes, Helper-Inducer
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Biological: Therapeutic vaccinations from A5058s — Participants will receive assigned interventions assigned in study A5058s.

SUMMARY:
The purpose of this study is to determine whether therapeutic HIV vaccines can help the immune system control HIV viral load after anti-HIV drugs are discontinued.

DETAILED DESCRIPTION:
This study is a rollover study for patients who participated in A5058s: Augmentation of HIV-Specific Helper and CTL Responses Through Therapeutic Vaccination in Individuals Receiving Potent Suppressive Antiretroviral Therapies. In A5058s, patients received a series of therapeutic vaccinations to elicit HIV-specific immune responses. This study will examine whether these vaccine-induced responses can control viral load in the absence of antiretroviral therapy (ART).

Upon study entry, patients will discontinue ART. During the first 6 weeks of the study, viral load will be monitored weekly and CD4+ T-cell counts will be monitored every other week. Viral load and CD4+ T-cell counts will be measured every other week from Week 6 through Week 24, then monthly until patients restart ART or until Week 48. Patients who reinitiate ART for any reason will be registered to Step 2 and followed for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participation in A5058s and receipt of a minimum of 7 sets of injections on that study
* Continuation of the same stable antiretroviral treatment that was given in A5058s for the last 3 months prior to A5172 entry, unless the regimen was changed for toxicity in the absence of virologic failure
* No less than 6 weeks and no more than 18 weeks since the last injection on A5058s prior to A5172 entry
* CD4+ T-cell count > 300 cells/mm3 obtained within 30 days prior to study entry
* HIV-1 RNA < 500 copies/ml obtained within 30 days prior to study entry
* Agreement to use approved methods of contraception

Exclusion Criteria:

* Pregnancy or breast-feeding
* Any of the following within 30 days prior to entry: acute infection requiring antibiotics, outbreak of herpes simplex virus (HSV) or herpes zoster, other acute medical illness, or surgery
* Symptomatic chronic infections other than HIV
* Malignancy that may require systemic therapy
* History of lymph node irradiation
* Use of immunoenhancing or immunosuppressive drugs within 30 days prior to entry, or any underlying disease of sufficient severity that these excluded drugs may be prescribed
* Hydroxyurea within 30 days prior to study entry
* Use of GM-CSF, G-CSF, M-CSF, IFN, IL-2, or other cytokines within 30 days prior to study entry
* Active drug or alcohol use or dependence that would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization until patient either completes therapy or is clinically stable on therapy for at least 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78
Dates: Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kalamus, M. D., Study Chair — Vanderbilt University Medical Center; Fred Valentine, M. D., Study Chair — NYU MEDICAL CENTER
Locations (14):
- United States (14):
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas

REFERENCES:
- [Background] Papasavvas E, Ortiz GM, Gross R, Sun J, Moore EC, Heymann JJ, Moonis M, Sandberg JK, Drohan LA, Gallagher B, Shull J, Nixon DF, Kostman JR, Montaner LJ. Enhancement of human immunodeficiency virus type 1-specific CD4 and CD8 T cell responses in chronically infected persons after temporary treatment interruption. J Infect Dis. 2000 Sep;182(3):766-75. doi: 10.1086/315748. Epub 2000 Aug 17. PMID 10950770
- [Background] Carcelain G, Tubiana R, Samri A, Calvez V, Delaugerre C, Agut H, Katlama C, Autran B. Transient mobilization of human immunodeficiency virus (HIV)-specific CD4 T-helper cells fails to control virus rebounds during intermittent antiretroviral therapy in chronic HIV type 1 infection. J Virol. 2001 Jan;75(1):234-41. doi: 10.1128/JVI.75.1.234-241.2001. PMID 11119593
- [Background] Deeks SG, Wrin T, Liegler T, Hoh R, Hayden M, Barbour JD, Hellmann NS, Petropoulos CJ, McCune JM, Hellerstein MK, Grant RM. Virologic and immunologic consequences of discontinuing combination antiretroviral-drug therapy in HIV-infected patients with detectable viremia. N Engl J Med. 2001 Feb 15;344(7):472-80. doi: 10.1056/NEJM200102153440702. PMID 11172188
- [Background] Ruiz L, Carcelain G, Martinez-Picado J, Frost S, Marfil S, Paredes R, Romeu J, Ferrer E, Morales-Lopetegi K, Autran B, Clotet B. HIV dynamics and T-cell immunity after three structured treatment interruptions in chronic HIV-1 infection. AIDS. 2001 Jun 15;15(9):F19-27. doi: 10.1097/00002030-200106150-00001. PMID 11416734
- [Background] Garcia F, Plana M, Vidal C, Cruceta A, O'Brien WA, Pantaleo G, Pumarola T, Gallart T, Miro JM, Gatell JM. Dynamics of viral load rebound and immunological changes after stopping effective antiretroviral therapy. AIDS. 1999 Jul 30;13(11):F79-86. doi: 10.1097/00002030-199907300-00002. PMID 10449278